CLINICAL TRIAL: NCT05363605
Title: A Phase 1/2 Study of [225Ac]-FPI-1966, [111In]-FPI-1967, and Vofatamab in Participants With FGFR3-expressing Advanced, Inoperable, Metastatic and/or Recurrent Solid Tumours
Brief Title: A Study of [225Ac]-FPI-1966 in Participants With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Fusion announced that it is discontinuing this study as part of a portfolio prioritization and assessment; Fusion no longer plans to pursue development of FPI-1966.
Sponsor: Fusion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FPI-1966-101
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor; Head and Neck Squamous Cell Carcinoma; Bladder Carcinoma; Susceptible FGFR3 Genetic Alterations; FGFR3; FGFR3 Overexpression; FGFR3 Receptor; FGFR3 Protein Overexpression; Ovarian Cancer; Colorectal Cancer; Breast Cancer; Liver Cancer; Lung Cancer; Gastric Cancer
Keywords: Actinium-225; Targeted Alpha Therapy; Radiopharmaceutical; Radioimmunoconjugate; Theranostic; Theragnostic; Radioligand; Antineoplastic agents; [225Ac]-FPI-1966
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Urinary Bladder Neoplasms; Ovarian Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Liver Neoplasms; Lung Neoplasms; Stomach Neoplasms | interventions — vofatamab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Depending on assigned cohort, [In111]-FPI-1967/[225Ac]-FPI-1966 will be administered with or without pre-dosing with vofatamab.
  Interventions: Drug: [225Ac]-FPI-1966; Drug: [111In]-FPI-1967; Biological: vofatamab
- Phase 2 (Experimental): Depending on assigned cohort, [In111]-FPI-1967/[225Ac]-FPI-1966 will be administered either with or without pre-administration of vofatamab, depending on the RP2D/regimen as determined in the phase 1 portion of the study.
  Interventions: Drug: [225Ac]-FPI-1966; Drug: [111In]-FPI-1967; Biological: vofatamab

INTERVENTIONS:
Drug: [225Ac]-FPI-1966 — [225Ac]-FPI-1966 is a targeted alpha therapeutic that consists of vofatamab, a bifunctional chelate, and actinium-225, an alpha particle emitting radionuclide. In Phase 1, the dose depends on cohort assignment. In Phase 2, the RP2D regimen will be administered.
Drug: [111In]-FPI-1967 — [111In]-FPI-1967 is an imaging agent that consists of vofatamab, a bifunctional chelate and indium-111 radionuclide. Participants will receive [111In]-FPI-1967 Injection of 185 MBq for imaging.
Biological: vofatamab — Vofatamab is a Fibroblast Growth Factor Receptor 3 (FGFR3)-targeting human monoclonal antibody without a radioisotope. In Phase 1, the dose depends on cohort assignment. In Phase 2, if pre-dosing with vofatamab is indicated, the RP2D regimen will be administered.

SUMMARY:
This first-in-human study evaluates safety, tolerability and distribution of [225Ac] FPI-1966, [111In]-FPI-1967, and vofatamab in patients with FGFR3-expressing solid tumors.

DETAILED DESCRIPTION:
In phase 1, cohort 1, the potential impact of pre-dose administration of vofatamab on the dosimetry, PK, safety, and tolerability of [225Ac]-FPI-1966 and [111In]-FPI-1967 will be evaluated.

In later phase 1 cohorts, [225Ac]-FPI-1966 will be evaluated at ascending dose levels. Participants will receive [111In]-FPI-1967 during the imaging screening period to assess FGFR3 expression and to determine biodistribution and estimate radiation exposure to critical organs.

Once the recommended phase 2 dose (RP2D) or regimen is established and confirmed, three tumour-agnostic expansion cohorts may be initiated in parallel.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed ICF prior to initiation of any study-specific procedures
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically and/or cytologically documented diagnosis of locally advanced, inoperable, or metastatic solid tumours
* Refractory to all standard treatments, or for whom standard treatment is not available, or tolerable, or is contraindicated, or the participant refuses standard therapy
* Measurable disease per RECIST v. 1.1
* Available tumour tissue (archival or fresh biopsy)
* Adequate bone marrow, heart, liver, and kidney function

Key Exclusion Criteria:

* Prior systemic radiopharmaceutical therapy within six months prior to the first dose of [111In]-FPI-1967
* Prior radiation therapy (RT) to bone marrow > 20 Gy
* RT within 30 days prior to the first dose of [111In]-FPI-1967
* Prior anti-cancer treatment (chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents) within a certain amount of time prior to administration of the first dose of [111In]-FPI-1967
* Concurrent serious co-morbidities that could limit participants' full participation and compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Phase 1: Phase 1: Incidence of AEs to evaluate safety and tolerability of [225Ac]-FPI-1966, [111In]-FPI-1967, and vofatamab. | Approximately 2 years post final administration
Phase 1: Maximum tolerated dose (MTD) of [225Ac]-FPI-1966 | Approximately 42 days post administration.
Phase 1: Radiation dose of [111In]-FPI-1967 and [225Ac]-FPI-1966 (whole body, organs, and selected regions of interest) | Within one week of administration
Phase 1: Effect of pre-dose administration of vofatamab on the radiation dosimetry of [111In]-FPI-1967 and [225Ac]-FPI-1966. | Within one week of administration
Phase 2: Objective response rate (ORR) (sum of complete and partial response) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | Up to two years post final administration.

SECONDARY OUTCOMES:
Phase 1 and 2: Anti-tumour activity of [225Ac]-FPI-1966 regimen measured by response per RECIST v1.1 | Approximately 2 years post final administration
Phase 1 and 2: Tumour uptake of [111In]-FPI-1967 by evaluating SPECT/CT and/or planar images | Within one week of administration
Phase 2: Radiation dose of [111In]-FPI-1967 and [225Ac]-FPI-1966 (whole body, organs, and selected regions of interest) | Within one week of administration
Phase 1 and 2: Clearance for radioactivity and for the targeting antibody. | 28 days post final [225Ac]-FPI-1966administration
Phase 1 and 2: Area under the curve (AUC) for radioactivity and targeting antibody | 28 days post final [225Ac]-FPI-1966administration.
Phase 1 and 2: Maximum concentration after dosing (Cmax) for radioactivity and targeting antibody. | 28 days post final[225Ac]-FPI-1966 administration
Phase 1 and 2: Half-life for radioactivity and targeting antibody. | 28 days post final [225Ac]-FPI-1966 administration
Phase 1: Changes in clearance for radioactivity and targeting antibody following pre-dose administration of vofatamab | 28 days post final [225Ac]-FPI-1966 administration
Phase 1: Changes in AUC for radioactivity and targeting antibody following pre-dose administration of vofatamab. | 28 days post final [225Ac]-FPI-1966 administration
Phase 1: Changes in Cmax for radioactivity and targeting antibody following pre-dose administration of vofatamab. | 28 days post final [225Ac]-FPI-1966 administration
Phase 1: Changes in half-life for radioactivity and targeting antibody following pre-dose administration of vofatamab | 28 days post final [225Ac]-FPI-1966 administration

CONTACTS AND LOCATIONS:
Overall Officials: Julia Kazakin, MD, Study Director — Fusion Pharmaceuticals Inc.
Locations (6):
- United States (4):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (2):
  - GC Murdoch, Murdoch, Western Australia
  - St Vincent's Hospital, Melbourne

REFERENCES:
- See also: Sponsor website — http://fusionpharma.com